CLINICAL TRIAL: NCT01840306
Title: Exosomal and Free Extracellular RNAs and Proteins as Predictive Biomarkers for HER2 Therapies in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 10-15
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; HER2 Positive Breast Cancer; HER2 Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: HER2 positive breast cancer: Female patients with newly diagnosed (including metastatic) HER2 positive breast cancer.
  Interventions: Other: Biomarker Analysis
- Cohort 2: HER2 negative breast cancer: Female patients with newly diagnosed HER2 negative breast cancer
  Interventions: Other: Biomarker Analysis

INTERVENTIONS:
Other: Biomarker Analysis

SUMMARY:
Primary Objective:

(i) To identify panels of RNAs and proteins predictive of response to HER2 targeted agents, considering clinical responses. (ii) To investigate associations between presence vs. absence (or relative levels) of identified extracellular (EC) RNAs/proteins and patients' clinicopathological characteristics, including age at diagnosis, time to progression and overall survival, as well as correlations with serum protein biomarkers routinely analysed for these patients. (iii) To compare HER2 positive samples versus HER2 negative samples for the existence of RNAs/proteins identified in (i) and (ii).

Secondary Objective:

To develop a predictive model for use in the HER2 positive population based on the most accurate and sensitive combination of the identified biomarkers.

DETAILED DESCRIPTION:
This is a translational pilot study, involving two patient cohorts, designed to identify predictive biomarkers for HER2 targeted therapy, which will be validated in a larger future study.

Cohort 1: 300 newly diagnosed (including metastatic) HER2 positive breast cancer patients. Cohort 2: 30 newly diagnosed HER2 negative breast cancer patients.

Blood specimens will be taken:

* before starting treatment (cohort 1 and 2)
* after receiving chemotherapy and before starting HER2 targeted treatment (if applicable) (cohort 1)
* within one month following 1st treatment of HER2 targeted treatment (cohort 1)
* approximately every 3 months (coinciding with formal disease assessment) while on HER2 targeted treatment for a maximum of 5 years (cohort 1)

Blood will be processed to serum, which will be analysed for RNA and protein biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a newly diagnosed (including metastatic) HER2 positive breast cancer, who is to commence HER2 targeted treatment.

   OR

   - Patient with a newly diagnosed HER2 negative breast cancer, who is to commence any type of treatment.
2. Patient must be female and aged 18 years or over.
3. Patient must provide written informed consent.

Exclusion Criteria:

1. Patients who do not fulfil the inclusion criteria mentioned above

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * HER2 positive breast cancer:Female patients with newly diagnosed (including metastatic) HER2 positive breast cancer.
  * HER2 negative breast cancer:Female patients with newly diagnosed HER2 negative breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2012-10-12 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Identification of Extra Cellular RNAs/proteins in sera from cancer patients | 7 years
  Identification of EC RNAs/proteins in sera from cancer patients, which correlate with their response to treatment

CONTACTS AND LOCATIONS:
Locations (11):
- Ireland (11):
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Letterkenny General Hospital, Donegal
  - Our Lady of Lourdes Hospital, Drogheda
  - Beacon Hospital, Dublin
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - The Adelaide & Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - Sligo General Hospital, Sligo
  - University Hospital Waterford, Waterford